CLINICAL TRIAL: NCT00153491
Title: Assessment of Adherence to a 6-Dose Regimen of Coartem for Treatment of Uncomplicated Malaria in Children Under 5 Years in Tanzania
Brief Title: Adherence to Lumefantrine-Artemether
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ifakara Health Research and Development Centre (Other)
Other Study IDs: CDC-NCID-3602
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Malaria, Uncomplicated
Keywords: malaria; artemether-lumefantrine; co-artem; Tanzania; adherence
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: artemether-lumefantrine

SUMMARY:
This is a study of how well caregivers of children with malaria adhere to the recommended regimen for lumefantrine-artemether (LA). Children were randomly assigned to either a group receiving directly observed treatment in hospital or to a group treated at home by the routine caregiver (typically, patient's mother). Clinical/parasitologic, hematologic, pharmacologic and qualitative parameters were monitored over a 28-day follow-up period and are used to evaluate drug adherence.

ELIGIBILITY:
Inclusion criteria:

* age < 5 years of age.
* axillary temperature >= 37.5oC
* unmixed infection with P. falciparum of between 1,000 and 250,000 asexual parasites/mm3 as determined by microscopic examination of thick, or thick and thin peripheral blood smears.
* parent/guardian's informed consent and willingness to participate in the study

Exclusion criteria:

* any evidence of severe or complicated malaria that would require hospitalization for treatment.
* reported allergy to any antimalarial drugs, including artemisinin derivatives and sulfa drugs.

Ages: 0 Years to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Start 2002-08; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Louise Causer, MBBS, MScPH, Study Director — Centers for Disease Control and Prevention; Salim Abdulla, MD, PhD, Study Director — Ifakara Health Research and Development Centre; Peter B Bloland, DVM, MPVM, Principal Investigator — Centers for Disease Control and Prevention; Stephen P Kachur, MD, MPH, Study Director — Centers for Disease Control and Prevention
Locations (1):
- Mkuranga District Hospital, Mkwanga, Mkuranga District, Tanzania